CLINICAL TRIAL: NCT00884793
Title: A Prospective Longitudinal Pilot Study to Measure the Effect of Intensification With Raltegravir +/- a Protease Inhibitor (PI) or Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) on HIV-1 Levels in the Gut
Brief Title: Pilot Study on the Effect of Adding Raltegravir +/- a Second Drug on HIV Levels in the Gut
Acronym: PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PLUS1
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Results first posted 2012-07-23 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: HIV; persistence; reservoirs; residual replication; gut; gut-associated lymphoid tissue; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; efavirenz; etravirine; Atazanavir Sulfate; fosamprenavir; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intensification with raltegravir +/- NNRTI or PI (Experimental): Intensification with raltegravir 400mg PO BID +/- a study PI or NNRTI
  Interventions: Drug: raltegravir; Drug: Study NNRTI; Drug: Study PI

INTERVENTIONS:
Drug: raltegravir — The baseline ART regimen will be intensified with raltegravir 400mg orally (PO) twice daily (BID) (all participants) +/- a study NNRTI or protease inhibitor (PI) (at the option of the participant and the study clinical team).
  Other Names: Isentress
Drug: Study NNRTI — Subjects who are not already on an NNRTI and who are suitable candidates will have the option of adding a study NNRTI (either efavirenz or etravirine).
  Other Names: efavirenz (Sustiva); etravirine (Intelence
Drug: Study PI — Subjects who are not on a PI and who are suitable candidates will have the option of adding a study PI. PIs used as study drugs will include atazanavir (+/- ritonavir), fosamprenavir (+/-ritonavir), lopinavir/ritonavir, and darunavir/ritonavir.
  Other Names: atazanavir (Reyataz, ATV); fosamprenavir (Lexiva, FPV, Telzir); lopinavir/ritonavir (Kaletra, LPV/r)

SUMMARY:
The "PLUS" study is a pilot study to measure the effect of therapy intensification (with raltegravir and optional second agent) on HIV levels in the gut and blood in patients on antiretroviral therapy (ART) with viral load < 50 copies/mL (herein referred to as "suppressed"). We hypothesize that there is ongoing replication in the gut despite suppressive ART and that this replication can be inhibited by the addition of one or two new antiretroviral drugs whose activity affects a distinct part of the viral life cycle. All study participants will have upper and lower endoscopy at baseline (before intensification) and after intensification. These endoscopies will be used to obtain gut tissue and single cells (for CD4+ cells) .

DETAILED DESCRIPTION:
The "PLUS" study is a prospective, longitudinal pilot study to measure the effect of therapy intensification (with raltegravir and possible addition of a study PI or NNRTI-Non-Nucleoside Reverse Transcriptase Inhibitor) on HIV-1 DNA/RNA levels in the gut-associated lymphoid tissue (GALT) and blood in patients on ART with viral load (VL) < 50 copies/mL (herein referred to as "suppressed"). We hypothesize that there is ongoing replication in the GALT despite suppressive ART and that this replication can be inhibited by the addition of one or two new antiretroviral drugs whose activity affects a distinct part of the viral life cycle. All study participants will have a colonoscopy and esophagogastroduodenoscopy (EGD) at baseline (before intensification) and a second colonoscopy with EGD 12 weeks after intensification. These endoscopies will be used to obtain GALT mononuclear cells (for CD4+ lymphocytes) as well as tissue for in situ hybridization and immunohistochemical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Infection with HIV-1, as documented by a licensed ELISA and confirmed by a Western blot or HIV-1 RNA at any time prior to study entry
3. On ART for at least 12 months prior to study entry with a regimen that includes at least two NRTIs and either an NNRTI or PI
4. No change in ART for at least 3 months prior to study entry.
5. CD4+ T cell count of 200 or greater within 30 days prior to study entry.
6. HIV-1 RNA level consistently below the limit of detection of commercial ultrasensitive assays (<50 copies/mL) for at least 6 months before study entry.
7. Women of reproductive potential (those who have not undergone surgical sterilization via hysterectomy, bilateral oophorectomy, or tubal ligation and who have had menses in the preceding 24 months) must have a negative urine or serum pregnancy test within 48 hours prior to study entry.
8. All subjects must agree not to participate in the process of conception (such as active attempts to impregnate or become pregnant, sperm or egg donation, in vitro fertilization) while receiving study drugs and for 6 weeks after stopping study drugs. If participating in sexual activity that could lead to pregnancy, the subject and/or partner should use at least two reliable methods of contraception, including oral contraceptive pills, an intrauterine device (IUD), condoms, and a diaphragm or cervical cap with spermicide.
9. Ability and willingness to provide informed consent.

Exclusion Criteria:

1. Any condition that, in the opinion of the GI specialist, would either be a contraindication to endoscopy or would increase the risk from sedation, endoscopy, or mucosal biopsies. These conditions may include, but are not limited to:

   * Significant complication (such as perforation) from prior endoscopy
   * Known bleeding diathesis
   * Platelet count < 100,000 per microliter
   * INR > 1.6
   * Current use of antiplatelet agents (aspirin, other NSAIDS, clopidogrel (Plavix), other antiplatelet agents) or anticoagulants (heparin, low molecular weight heparin, warfarin, lepirudin, or other anticoagulants) and inability to temporarily hold such medications for endoscopy.
   * Active angina, unstable angina, or MI within 2 months prior to study entry
   * Decompensated CHF
   * Respiratory insufficiency with FEV1 < 1L, resting hemoglobin saturation of <92%, or need for oxygen supplementation
   * OSA requiring CPAP
   * Ongoing substance abuse
   * Peripheral glucose > 350 mg/dL
2. Prior use of raltegravir
3. Any condition that, in the opinion of the infectious disease (ID) specialist, would be a contraindication to raltegravir. These conditions may include, but are not limited to: unstable clinical condition (such as recent hospitalization, cancer with need for chemotherapy or radiation); severe hepatic insufficiency; need for contraindicated medicines; breastfeeding; or high risk for myopathy or rhabdomyolysis.
4. Calculated creatinine clearance (CrCl) < 50 mL/min, as estimated by the Cockcroft-Gault equation
5. AST (SGOT), ALT (SGPT), alkaline phosphatase, or bilirubin > 3x the upper limit of normal (ULN).
6. LDL > 200 mg/dL or TG > 400 mg/dL in fasting lipids, as measured within three months prior to screening or at the time of screening
7. Plan to change the background ART within 16 weeks after study entry
8. Receipt of any HIV vaccine
9. Receipt of a non-HIV vaccine within 30 days prior to study entry
10. An opportunistic infection within 60 days prior to study entry
11. Use of significant immunosuppressive medications (such as systemic corticosteroids, tacrolimus, sirolimus, mycophenolate, azathioprine, interferon, and cancer chemotherapy) within 60 days prior to study entry.
12. Active drug or alcohol abuse that, in the opinion of the investigator, would interfere with adherence to the requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, MD, Principal Investigator — San Francisco General Hospital (SFGH) and University of California San Francisco (UCSF); Joseph K Wong, MD, Principal Investigator — San Francisco VA Medical Center (SFVAMC) and University of California, San Francisco (UCSF); Steven Yukl, MD, Principal Investigator — SFVMAC and UCSF
Locations (2):
- United States (2):
  - San Francisco General Hospital, San Francisco, California
  - San Francisco VA Medical Center (SFVAMC), San Francisco, California

REFERENCES:
- [Result] Yukl SA, Gianella S, Sinclair E, Epling L, Li Q, Duan L, Choi AL, Girling V, Ho T, Li P, Fujimoto K, Lampiris H, Hare CB, Pandori M, Haase AT, Gunthard HF, Fischer M, Shergill AK, McQuaid K, Havlir DV, Wong JK. Differences in HIV burden and immune activation within the gut of HIV-positive patients receiving suppressive antiretroviral therapy. J Infect Dis. 2010 Nov 15;202(10):1553-61. doi: 10.1086/656722. Epub 2010 Oct 12. PMID 20939732
- [Result] Yukl SA, Shergill AK, McQuaid K, Gianella S, Lampiris H, Hare CB, Pandori M, Sinclair E, Gunthard HF, Fischer M, Wong JK, Havlir DV. Effect of raltegravir-containing intensification on HIV burden and T-cell activation in multiple gut sites of HIV-positive adults on suppressive antiretroviral therapy. AIDS. 2010 Oct 23;24(16):2451-60. doi: 10.1097/QAD.0b013e32833ef7bb. PMID 20827162

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensification Arm: In addition to continuing the baseline ART regimen (2 NRTIs and either a PI or NNRTI), all subjects will receive raltegravir 400mg PO (by mouth) BID (twice daily). Subjects who are suitable candidates will have the option of adding a second drug, consisting of either a study NNRTI or a study PI. Subjects who are not already on an NNRTI and who are suitable candidates will have the option of adding a study NNRTI (either efavirenz or etravirine), while subjects who are not on a PI and who are suitable candidates will have the option of adding a study PI. PIs used as study drugs will include atazanavir (+/- ritonavir), fosamprenavir (+/-ritonavir), lopinavir/ritonavir, and darunavir/ritonavir.
Period: Overall Study
Arm/Group | Intensification Arm
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intensification Arm
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Had a Decrease in HIV RNA Per Million CD4+ T Cells in the Ileum
Description: Number of subjects who had a decrease from week 0 to week 12 in unspliced cell-associated HIV RNA per million CD4+ T cells in the ileum
Time Frame: 12 weeks
Population: We analyzed data from all subjects who had endosocopies at week 12.
Measure: Number; unit: participants
Groups:
- Intensification Arm: 5 subjects were intensified with raltegravir alone, 2 received raltegravir plus efavirenz, and 1 received raltegravir plus ritonavir/darunavir
Arm/Group | Intensification Arm
Number analyzed (Participants) | 7
participants | 5

2. Secondary Outcome: Number of Subjects Who Experienced an Increase in CD4+ T Cells (as a % of All Cells) in the Ileum.
Description: Number of subjects who experienced an increase in CD4+ T cells (as a % of all cells) in the ileum (by flow cytometry) from week 0 to week 12.
Time Frame: 12 weeks
Population: Includes all with gut samples from week 12.
Measure: Number; unit: participants
Arm/Group | Intensification Arm
Number analyzed (Participants) | 7
participants | 6

3. Secondary Outcome: Number of Subjects Who Experienced an Increase in CD4% in the Ileum.
Description: Number of subjects who experienced an increase from week 0 to week 12 in CD4+ T cells (as a % of T cells, by flow cytometry) in the ileum
Time Frame: 12 weeks
Population: Includes all those who had endoscopy at week 12
Measure: Number; unit: participants
Arm/Group | Intensification Arm
Number analyzed (Participants) | 7
participants | 5

4. Secondary Outcome: Average Change in "Activated" (CD38+HLADR+) CD8+ T Cells in the Ileum
Description: Average of changes(week 0-week 12) in the % of CD8+ T cells that are CD38+HLA-DR+, by flow cytometry
Time Frame: 12 weeks
Population: All patients who had endoscopy at week 12.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Intensification Arm
Number analyzed (Participants) | 7
percentage change | -5.4 (4.5)

ADVERSE EVENTS:
Time Frame: 12 weeks of intensification with raltegravir, followed by cessation of raltegravir (but not baseline ART) and monitoring for an additional 4 weeks
Arm/Group | Intensification Arm
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
1) relatively small number of participants; 2) intensification may have been too short; 3)the biopsies themselves can cause inflammation/microbial leakage; 4) sampling may miss viral replication if it occurs in temporally and spatially-discrete foci

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes